CLINICAL TRIAL: NCT04950244
Title: Diagnostic Evaluation of Out-of-hospital High-sensitivity Troponin I in Patients Presenting Chest Pain
Acronym: VALIDATE
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VALIDATE
Record Dates: First submitted 2021-06-22; First posted 2021-07-06 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2023-01

CONDITIONS: Chest Pain
Keywords: High-sensitivity cardiac Troponin I; Troponin I HS
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High-sensitivity cardiac troponin I (hs-cTnI) — Capillary and veinous whole blood sampling for hs-cTnI was collected. The sample was tested at the bedside with a point-of-care device (Atellica VTLi, Siemens Healthineers).
  The result of both hs-c TnI values obtained was blinded to the treating physician

SUMMARY:
Conducting an analysis of the clinical performance of high-sensitivity cardiac troponin I, tested in the out-of-hospital setting, for ruling out cardiac origin in acute onset chest pain.

Acute onset chest pain is a complex symptom to narrow down in the out-of-hospital setting. This is due to the difficulty of obtaining pertinent information over the phone, and the absence of validated dispatch scores or criteria.

In France, the current standard of care relies on the rapid dispatch of Emergency Medical Response Teams along with a physician in patients presenting symptoms evocative of Coronary Artery Disease or Myocardial Infarction.

Typical anginal pain includes retrosternal pressure pain radiating to the jaw, neck, or left arm. Diagnostic work-up includes anamnesis, physical examination, routine blood work, and ECG.

In the absence of signification ST-segment modifications, the gold standard relies on trending serum Troponin T and I in the hospital setting .

This study aims to analyze the clinical performance of high-sensitivity cardiac Troponin I assays (hs-cTnI) in the out-of-hospital setting using a point-of-care device ; Atellica VTLi (Siemens Healthineers)

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Presenting with evocative acute onset chest pain

Exclusion Criteria:

* ECG modifications with ST segment elevations
* Patients for whom anginal origin was excluded in the out-of-hospital setting
* Medical evaluation in a delay inferior to 20 minutes
* Patients without medical insurance
* Pregnant or lactating women
* Patients under reinforced guardianship, minors, patients in hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: overall population of callers to the emergency dispatch center
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Clinical performance of hs-cTnI for rule-out of cardiac origin of chest pain in the out of hospital setting | 3 hours
  Determining the more appropriate cut off in terms of specificity and sensitivity to rule out chest pain in relation to coronary artery disease, based on the ROC curve.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT04950244/SAP_000.pdf